CLINICAL TRIAL: NCT05237427
Title: Determination of Respiratory Muscle Endurance in Healthy Adult Individuals
Brief Title: Inspiratory Muscle Endurance of Adults
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Selda GOKCEN, Lecturer, Kutahya Health Sciences University
Other Study IDs: 100
Record Dates: First submitted 2022-01-18; First posted 2022-02-14 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the reference value ranges for healthy adults of the incremental threshold load test, which evaluates respiratory muscle endurance.

DETAILED DESCRIPTION:
Since respiratory muscles are used in daily life at the submaximal level, evaluation of their endurance is more meaningful functionally. In addition, evaluation of endurance with respiratory muscle strength is effective in determining respiratory muscle dysfunction. Failure to routinely evaluate respiratory muscle endurance, which is one of the main components of respiratory muscle function, may lead to failure to identify respiratory muscle dysfunction in early stage respiratory patients who have not yet developed muscle strength loss. However, normal value ranges have not been determined for the respiratory muscle endurance test.

Determining the normal value ranges for this test will help determine muscle fatigue and investigate the physiological course in respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Not having any disease
* Not exercising regularly
* Not smoking

Exclusion Criteria:

* Having a respiratory disease
* Have heart disease
* Have a neuromuscular disease
* Have Scoliosis
* Having had thoracic surgery
* Having experienced the respiratory muscle endurance protocol before

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers between the ages of 18-35
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Incremental threshold loading test. | 15 minute
  A measure of endurance of inspiratory muscles.
Maximal inspiratory pressure | 20 minute
  A measure of the strength of inspiratory muscles

SECONDARY OUTCOMES:
Pulmonary function test - Forced expiratory volume in 1 second (FEV1) | 5 minute
  The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration. It is lung function test that are measured during spirometry. This pulmonary function test measurements were made to confirm that the respiratory function parameters of the participants were within the normal range. .
Pulmonary function test - Forced vital capacity (FVC) | 5 minute
  Forced vital capacity (FVC) is lung function test that are measured during spirometry. This pulmonary function test measurement is applied to confirm that the respiratory function parameters of the participants were within the normal range.
Maximal voluntary ventilation (MVV) | 5 minute
  It is a test that measures inspiratory endurance. MVV is the largest amount of air that a person can inhale and then exhale during a 12- to 15-s interval with maximal voluntary effort. It is determined by spirometry measurement.
International Physical Activity Questionnaire - Short Form | 5 minute
  This questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in the metabolic equivalent of task (MET)-minute/week and time spent sitting.

OTHER OUTCOMES:
Anthropometric assessment | 5 minute
  Body weight was assessed with a digital scale in the orthostatic position, without shoes, with minimal clothing. Height was measured with the feet parallel and adjacent to each other, the arms extended by the body, and the head in a neutral position. Correlations between inspiratory muscle endurance of the incremental threshold loading protocol and anthropometric characteristics will be shown.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Gokcen, Principal Investigator — Kutahya Health Sciences University; Ozgen Aras, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)